CLINICAL TRIAL: NCT04958668
Title: Prospective Evaluation of Volatile Sedation With Regard to Awakening Behaviour and Extubation Capacity in Patients Undergoing Heart Valve Surgery
Brief Title: Prospective Evaluation of Volatile Sedation After Heart Valve Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Goethe University (Other)
Responsible Party: Principal Investigator, Armin N. Flinspach, Principal Investigator, Goethe University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: 20-1050
Record Dates: First submitted 2021-06-28; First posted 2021-07-12 (Actual); Last update posted 2024-01-09 (Actual); Status verified 2024-01

CONDITIONS: Valve Heart Disease; Awakening Early
MeSH Terms: conditions — Heart Valve Diseases; Sleep Initiation and Maintenance Disorders

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Volatile procedere (Active Comparator): Intensive care treatment with demand-adapted sedation with volatile anaesthetics
  Interventions: Other: Post-operative intensive care using volatile sedation
- Conventional procedere (No Intervention): Conventional Intensive care treatment with demand-adapted sedation with intravenous sedatives

INTERVENTIONS:
Other: Post-operative intensive care using volatile sedation — Patients admitted after valve surgery are receiving intensive care using volatile sedative per anaesthetic conserving device. The subject of the study is medical and nursing time management..
  Arms: Volatile procedere

SUMMARY:
Cardiac surgery is a complex operative procedure with a substantial risk of postoperative complications, so that patients undergoing valve surgery are usually transferred to the intensive care unit postoperatively. Various substances are used to maintain the required sedation, such as volatile anaesthetics and intravenous sedatives combined with analgetic therapy using opioids.

The study intends to investigate to what extent the already well-described effect of volatile anaesthetics on recovery can be realised despite the need for differentiated intensive care and medical management.

ELIGIBILITY:
Inclusion Criteria:

* Valve reconstruction or valve replacement
* Must be capable to giving written consent

Exclusion Criteria:

* Intolerance to volatile anaesthetics (e.g. malignant hyperthermia)
* Severe obstructive pulmonary disease
* Extended aortic arch or ascending aorta surgery
* Age <18 years

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2021-11-01 (Actual); Primary Completion 2023-08-28 (Actual); Study Completion 2023-12-01 (Actual)

PRIMARY OUTCOMES:
Time to extubation | through study completion, an average of 2 days
  Time from admission on ICU until awakening and Extubation.

SECONDARY OUTCOMES:
Time to neurocognitive assessability | through study completion, an average of 2 days
  Time from admission on ICU until awake and neurocognitive assessable.
Required setup time of the intensive care workplace | through study completion, up to 24 hours
  Required setup time of the intensive care workplace to provide volatile or intravenous sedation.
Factor related to the course of intensive care: blood loss | through study completion, an average of 24 hours
  Measured Postoperative Blood Loss
Factor related to the course of intensive care: kidney injury | through study completion, an average of 24 hours
  Measured increases in serum renal retention levels: creatinine and urea in terms of renal failure according to Kidney Disease - Improving Global Outcomes (KDIGO) criteria.
Factor related to the course of intensive care: acid-base balance | through study completion, an average of 24 hours
  Measured serum lactate levels and hypercapnia
Factor related to the course of intensive care: lung function parameters | through study completion, an average of 24 hours
  Required inspiratory oxygen fraction
Factor related to the course of intensive care:cardiovascular medication | through study completion, an average of 24 hours
  Required dosage of adrenaline, noradrenaline, vasopressin or milrinone
Factors related to the course of operative procedure | through study completion, up to 24 hours
  time of the intraoperative procedure including the heart-lung-machine
Intra-hospital mortality | through study completion, an average of 7 days
  Intra-hospital mortality - Safety outcome
Liver failure | through study completion, an average of 7 days
  Intra-hospital liver failure - Safety outcome
postoperative nausea and vomiting | through study completion, up to 24 hours
  Detection of postoperative nausea and vomiting

CONTACTS AND LOCATIONS:
Overall Officials: Armin N Flinspach, M.D., Principal Investigator — JWGoethe University
Locations (1):
- University Hospital Frankfurt, Frankfurt am Main, Hesse, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Flinspach AN, Raimann FJ, Kaiser P, Pfaff M, Zacharowski K, Neef V, Adam EH. Volatile versus propofol sedation after cardiac valve surgery: a single-center prospective randomized controlled trial. Crit Care. 2024 Apr 5;28(1):111. doi: 10.1186/s13054-024-04899-y. PMID 38581030
- [Derived] Flinspach AN, Herrmann E, Raimann FJ, Zacharowski K, Adam EH. Evaluation of volatile sedation in the postoperative intensive care of patients recovering from heart valve surgery: protocol for a randomised, controlled, monocentre trial. BMJ Open. 2022 Feb 23;12(2):e057804. doi: 10.1136/bmjopen-2021-057804. PMID 35197356